CLINICAL TRIAL: NCT05039762
Title: Intracorporeal vs. Extracorporeal Anastomosis in Patients Undergoing Laparoscopic Right Hemicolectomy for Colonic Cancer - A Prospective Cohort Study
Brief Title: Intracorporeal vs. Extracorporeal Anastomosis in Patients Undergoing Laparoscopic Right Hemicolectomy for Colonic Cancer
Acronym: ICEA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Benedicte Schelde-Olesen, Principal investigator, University of Southern Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICEA-051-2016-NQ
Record Dates: First submitted 2020-11-11; First posted 2021-09-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Colon Cancer
Keywords: Laparoscopic right hemicolectomy; Intracorporeal anastomosis; Extracorporeal anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single center, non-randomized, non-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal anastomosis (Active Comparator): Laparoscopic right hemicolectomy with Extracorporeal anastomosis in patients with colon cancer.
  Interventions: Procedure: Extracorporeal anastomosis
- Intracorporeal anastomosis (Experimental): Laparoscopic right hemicolectomy with Intracorporeal anastomosis in patients with colon cancer.
  Interventions: Procedure: Intracorporeal anastomosis

INTERVENTIONS:
Procedure: Extracorporeal anastomosis — Laparoscopic right hemicolectomy will be carried out. The dissection is performed laparoscopically. When the right hemicolon is sufficiently mobilized and the vessels (ileocolic pedicle, right colic pedicle and the right branch of the middle colic pedicle) are ligated, a horizontal incision in the upper right quadrant is made. Through this incision the right hemicolon is extracted, the small bowel and the transverse colon are divided using staplers. The side-to-side ileocolic anastomosis is then handsewn.
  Arms: Extracorporeal anastomosis
Procedure: Intracorporeal anastomosis — Laparoscopic right hemicolectomy will be carried out. The dissection is performed laparoscopically. The right hemicolon is mobilized and the vessels (ileocolic pedicle, right colic pedicle and the right branch of the middle colic pedicle) are ligated. The small bowel and the transverse colon are then divided using laparoscopic staplers. The side-to-side ileocolic anastomosis is formed by creating a small opening in the small bowel and the transverse colon, through which the laparoscopic stapler is used to join the bowel ends. The remaining opening is sutured laparoscopically. The specimen is retrieved through a Pfannenstiel incision.
  Arms: Intracorporeal anastomosis

SUMMARY:
In this study, the investigators will compare extracorporeal anastomosis (EA) with intracorporeal anastomosis (IA) in patients undergoing elective laparoscopic hemicolectomy for right colon cancer.

DETAILED DESCRIPTION:
At Odense University Hospital, Svendborg, current standard treatment for right colon cancer is laparoscopic hemicolectomy with extracorporeal anastomosis (EA).

To reduce the risk of adverse events, such as fascial dehiscence and later development of incisional hernia, right hemicolectomy with intracorporeal anastomosis has been introduced.

When performing a laparoscopic right hemicolectomy the dissection is carried out intracorporeally and the transection and anastomosis is made extracorporeally (EA technique). For IA technique the cancer bearing segment is resected and the bowel ends joined intracorporeally with laparoscopic technique, and the specimen is then retrieved through a Pfannenstiel incision.

Previous series have shown shorter hospital stay as well as shorter time to bowel recovery in patients treated with IA compared to EA, without increasing the risk of severe complications or compromising the oncological outcome.

The aim of this study is to investigate whether IA in patients undergoing right hemicolectomy reduces the overall complication rate compared to EA evaluated by Comprehensive Complication Index (CCI) .

51 patients will be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with right colon cancer
* Eligible for elective laparoscopic right hemicolectomy with primary anastomosis.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* CT staged T1-T3M0 tumour.

Exclusion Criteria:

* Pregnancy
* Mental incompetence
* Acute right hemicolectomy before the intended elective surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall complication rate | 30 days
  According to the Comprehensive Complication Index (CCI) based on the Clavien Dindo classification of postsurgical complications.
  CCI is a continuous scale from 0-100 (0 equals no complications, 100 equals death)

SECONDARY OUTCOMES:
Surgical stress response | Up to 30 days
  Evaluated by C-reactive protein (CRP), leucocytes and National Early Warning Score (NEWS).
  NEWS is an aggregate scoring system, based on physiological measurements, designed to help detect acute illness. Minimum score of 0 indicates normal measurements. The score increases with further deviation from the norm, with a maximum score of 20.
Time until bowel recovery | Up to 30 days
  Measured in hours from end of surgery to first flatus and first bowel movement respectively
Length of hospital stay | Up to 30 days
  Measured in hours from end of surgery until the patient is discharged
Postoperative pain | Up to 30 days
  Registered daily using Visual analogue scale (VAS) for pain. The scale ranging from 0-10, 0 being no pain, 10 being worst pain imaginable.
Hernia rate | 3 years
  Based on CT scans 1 and 3 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Benedicte Schelde-Olesen, MD, Principal Investigator — Odense University Hospital, Svendborg
Locations (1):
- Odense University Hospital, Svendborg, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwenk W, Haase O, Neudecker J, Muller JM. Short term benefits for laparoscopic colorectal resection. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003145. doi: 10.1002/14651858.CD003145.pub2. PMID 16034888
- [Background] Ricci C, Casadei R, Alagna V, Zani E, Taffurelli G, Pacilio CA, Minni F. A critical and comprehensive systematic review and meta-analysis of studies comparing intracorporeal and extracorporeal anastomosis in laparoscopic right hemicolectomy. Langenbecks Arch Surg. 2017 May;402(3):417-427. doi: 10.1007/s00423-016-1509-x. Epub 2016 Sep 5. PMID 27595589
- [Background] Wu Q, Jin C, Hu T, Wei M, Wang Z. Intracorporeal Versus Extracorporeal Anastomosis in Laparoscopic Right Colectomy: A Systematic Review and Meta-Analysis. J Laparoendosc Adv Surg Tech A. 2017 Apr;27(4):348-357. doi: 10.1089/lap.2016.0485. Epub 2016 Oct 21. PMID 27768552
- [Background] van Oostendorp S, Elfrink A, Borstlap W, Schoonmade L, Sietses C, Meijerink J, Tuynman J. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Jan;31(1):64-77. doi: 10.1007/s00464-016-4982-y. Epub 2016 Jun 10. PMID 27287905
- [Background] Vergis AS, Steigerwald SN, Bhojani FD, Sullivan PA, Hardy KM. Laparoscopic right hemicolectomy with intracorporeal versus extracorporeal anastamosis: a comparison of short-term outcomes. Can J Surg. 2015 Feb;58(1):63-8. doi: 10.1503/cjs.001914. PMID 25621913
- [Background] Hellan M, Anderson C, Pigazzi A. Extracorporeal versus intracorporeal anastomosis for laparoscopic right hemicolectomy. JSLS. 2009 Jul-Sep;13(3):312-7. PMID 19793468
- [Background] Grams J, Tong W, Greenstein AJ, Salky B. Comparison of intracorporeal versus extracorporeal anastomosis in laparoscopic-assisted hemicolectomy. Surg Endosc. 2010 Aug;24(8):1886-91. doi: 10.1007/s00464-009-0865-9. Epub 2010 Jan 29. PMID 20112118
- [Background] Milone M, Elmore U, Di Salvo E, Delrio P, Bucci L, Ferulano GP, Napolitano C, Angiolini MR, Bracale U, Clemente M, D'ambra M, Luglio G, Musella M, Pace U, Rosati R, Milone F. Intracorporeal versus extracorporeal anastomosis. Results from a multicentre comparative study on 512 right-sided colorectal cancers. Surg Endosc. 2015 Aug;29(8):2314-20. doi: 10.1007/s00464-014-3950-7. Epub 2014 Nov 21. PMID 25414066
- [Background] Emile SH, Elfeki H, Shalaby M, Sakr A, Bassuni M, Christensen P, Wexner SD. Intracorporeal versus extracorporeal anastomosis in minimally invasive right colectomy: an updated systematic review and meta-analysis. Tech Coloproctol. 2019 Nov;23(11):1023-1035. doi: 10.1007/s10151-019-02079-7. Epub 2019 Oct 23. PMID 31646396
- [Background] Bollo J, Turrado V, Rabal A, Carrillo E, Gich I, Martinez MC, Hernandez P, Targarona E. Randomized clinical trial of intracorporeal versus extracorporeal anastomosis in laparoscopic right colectomy (IEA trial). Br J Surg. 2020 Mar;107(4):364-372. doi: 10.1002/bjs.11389. Epub 2019 Dec 17. PMID 31846067
- [Background] Mari GM, Crippa J, Costanzi ATM, Pellegrino R, Siracusa C, Berardi V, Maggioni D. Intracorporeal Anastomosis Reduces Surgical Stress Response in Laparoscopic Right Hemicolectomy: A Prospective Randomized Trial. Surg Laparosc Endosc Percutan Tech. 2018 Apr;28(2):77-81. doi: 10.1097/SLE.0000000000000506. PMID 29360701
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Petersen JA. Early warning score challenges and opportunities in the care of deteriorating patients . Dan Med J. 2018 Feb;65(2):B5439. PMID 29393044
- [Background] Williams B. The National Early Warning Score and the acutely confused patient. Clin Med (Lond). 2019 Mar;19(2):190-191. doi: 10.7861/clinmedicine.19-2-190. No abstract available. PMID 30872312
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Derived] Hougaard ES, Schelde-Olesen B, Al-Najami I, Buchbjerg T, Rasmussen BSB, Bugge L, Kolbro T, Moller S, Ellebaek MB. Short-term outcomes for intracorporeal vs. extracorporeal anastomosis in laparoscopic right hemicolectomy for colonic cancer-a prospective cohort study (ICEA-study). Int J Colorectal Dis. 2025 Apr 8;40(1):90. doi: 10.1007/s00384-025-04882-1. PMID 40198370